CLINICAL TRIAL: NCT05885217
Title: Evaluation of Serum MicroRNA in Acne Vulgaris and Relation to Acne Severity
Brief Title: Measurement of Serum microRNA in Acne Vulgaris Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Alshayma Gamal Fouad, doctor, South Valley University
Other Study IDs: serum microRNA
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1: mild form of acne vulgaris
  Interventions: Other: measure serum MicroRNA in acne vulgaris
- group2: moderate form of acne vulgaris
  Interventions: Other: measure serum MicroRNA in acne vulgaris
- group 3: severe form of acne vulgaris
  Interventions: Other: measure serum MicroRNA in acne vulgaris
- group 4: control group
  Interventions: Other: measure serum MicroRNA in acne vulgaris

INTERVENTIONS:
Other: measure serum MicroRNA in acne vulgaris — Quantitively assay of serum microRNA level will be measured control by performing an enzyme-linked immune sorbent assay (E LISA)

SUMMARY:
The aim of the study is to:

1. Evaluation of serum microRNA in acne vulgaris and compare to control group
2. Evaluate correlation with acne vulgaris severity

DETAILED DESCRIPTION:
Acne vulgaris is a common chronic skin disease involving blockage and inflammation of pilosebaceous units.

Acne vulgaris is characterized by non-inflammatory, open or closed comedones and by Inflammatory lesions include papules, pustules and nodules. Affecting mostly the face but also the back and chest.

Acne vulgaris may have a psychological impact on any patient, regardless of the severity or the grade of the disease.

Prevalence of self-reported acne was 34.7%. Females significantly reported acne more frequently than males (39.1% vs. 30.3%) Prevalence of clinically confirmed acne was 24.4%, with higher rates among females (28.6%) than males (20.2%).(4) the pathogenesis result from increased sebum production (due to increased activity of androgens and (IGF-1), excessive deposition of keratin in pilosebaceous follicles leading to comedo formation, colonization of the follicle by Propionibacterium acnes bacteria, and the local release of pro-inflammatory chemicals in the skin through certain inflammatory mechanisms.

recently, Inflammation is a key feature in the pathogenesis of acne vulgaris , with various chemokines and cytokines that contribute to fuel a vicious cycle.

In addition, genetics is also a key factor in the pathophysiology of acne. MicroRNAs(MiRNAs) are a class of endogenous, short (19-23 nucleotides in length), which regulate the expression of genes via translational repression or degradation of target messenger RNAs.Recently, the role of miRNAs has also been reviewed for the pathogenesis of various inflammatory skin conditions such as psoriasis, eczema, atopic dermatitis and toxic epidermal necrolysis.

MiRNAs are present not only in the intracellular space, but also in extracellular spaces such as serum, urine, and saliva. This study is the first to evaluate microRNA in serum of acne vulgaris patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy persons of both sexes with mild, moderate and severe acne vulgaris.
* 2. Patients with acne vulgaris not receiving any topical or systemic treatments for acne at least 6 months

Exclusion Criteria:

* 1. Pregnant and lactating women
* 2. Patients with history of cardiovascular disorder, renal disease, malignancy, chronic liver disease
* 3. Patients with history of depression or mental illness
* 4. Diabetes type 2
* 5. Obesity
* 6. Patient with history of melasma, psoriasis, eczema, atopic dermatitis and toxic epidermal necrolysis.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the study will include patients with active acne vulgaris ( mild, moderate, severe) who will come to the out-patient dermatologic clinic and match inclusion & exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate serum levels of microRNA in acne vulgaris patients | baseline
  Evaluate serum levels of microRNA in acne vulgaris patients and compare with levels in healthy controls and determine correlation with acne severity

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mohammed Ibrahim, professor, Study Director — South Valley University; Abdulrahman Abdul Hamid Alsaied, professor, Study Director — South Valley University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hazarika N. Acne vulgaris: new evidence in pathogenesis and future modalities of treatment. J Dermatolog Treat. 2021 May;32(3):277-285. doi: 10.1080/09546634.2019.1654075. Epub 2019 Aug 29. PMID 31393195
- [Background] Kellett SC, Gawkrodger DJ. The psychological and emotional impact of acne and the effect of treatment with isotretinoin. Br J Dermatol. 1999 Feb;140(2):273-82. doi: 10.1046/j.1365-2133.1999.02662.x. PMID 10233222
- [Background] Tayel K, Attia M, Agamia N, Fadl N. Acne vulgaris: prevalence, severity, and impact on quality of life and self-esteem among Egyptian adolescents. J Egypt Public Health Assoc. 2020 Nov 5;95(1):30. doi: 10.1186/s42506-020-00056-9. PMID 33165744
- [Background] Goulden V, McGeown CH, Cunliffe WJ. The familial risk of adult acne: a comparison between first-degree relatives of affected and unaffected individuals. Br J Dermatol. 1999 Aug;141(2):297-300. doi: 10.1046/j.1365-2133.1999.02979.x. PMID 10468803
- [Background] Borgia F, Peterle L, Custurone P, Vaccaro M, Pioggia G, Gangemi S. MicroRNA Cross-Involvement in Acne Vulgaris and Hidradenitis Suppurativa: A Literature Review. Int J Mol Sci. 2022 Mar 17;23(6):3241. doi: 10.3390/ijms23063241. PMID 35328662
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- See also: Mstfa S A G. An Overview About Acne Vulgaris. Journal of Pharmaceutical Negative Results.(2022):4395-4402 — https://scholar.google.com/scholar?hl=ar&as_sdt=0%2C5&q=2.%09Mustafa+S+A+G.+An+Overview+About+Acne+Vulgaris.+Journal+of+Pharmaceutical+Negative+Results.%282022%29%3A4395-4402+&btnG=
- See also: U.S. Department of Health and Human Services Food and Drug Administration Center for Drug Evaluation and Research (CDER).Guidance for industry. Acne vulgaris: developing drugs for treatment.(2005). — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/acne-vulgaris-establishing-effectiveness-drugs-intended-treatment